CLINICAL TRIAL: NCT01221922
Title: A Study of the RevLite Q-Switched Neodymium: Yttrium-Aluminum-Garnet (Nd:YAG) Laser for the Treatment of Acne Scars in Fitzpatrick Skin Types III-VI
Brief Title: Laser Treatment of Acne Scars in Fitzpatrick Skin Types III-VI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ConBio, a Cynosure Company (Industry)
Responsible Party: Sponsor
Organization: Cynosure, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C67-10-A
Record Dates: First submitted 2010-10-14; First posted 2010-10-18 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-11

CONDITIONS: Acne Scars

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acne treatment (Experimental): Treatment of acne scars
  Interventions: Device: RevLite Q-Switched Nd:YAG Laser

INTERVENTIONS:
Device: RevLite Q-Switched Nd:YAG Laser — Laser treatment once every 2 weeks for a total of 10 treatments.

SUMMARY:
The purpose of this study is to evaluate the RevLite Q-Switched Neodymium: Yttrium-Aluminum-Garnet (Nd:YAG) Laser in the treatment of acne scars in darker skin types (Fitzpatrick Skin Types III, IV, V and VI).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older with Fitzpatrick Skin Type III, IV, V or VI
* Evidence of atrophic scarring

Exclusion Criteria:

* Pregnancy, lactating or planning to become pregnant during the study
* History of cutaneous photosensitization, porphyria, and hypersensitivity to porphyrins or photodermatosis
* Any skin pathology or condition that could interfere with the evaluation or requires the use of interfering topical or systemic therapy
* Any condition which, in the investigator's opinion, would make it unsafe for the subject to participate
* Currently enrolled in an investigational drug or device trial, or has received an investigational drug or been treated with an investigational device within 30 days prior to entering the study
* Subject is unable to communicate or cooperate with the investigator due to language problems, poor mental development, or impaired cerebral function
* Subject may be unreliable for the study. This includes subjects who engage in excessive alcohol intake or drug abuse, or subjects who are unable to return for scheduled follow-up visits
* Use of oral or topical isotretinoin therapy within 6 months prior to enrollment. With the exception of isotretinoin, subjects will be allowed to continue their topical or oral acne medications during the trial
* Need to be exposed to artificial tanning devices or excessive sunlight during the trial
* Prior treatment with parenteral gold therapy
* Diabetes Type I or II, Lupus, Scleroderma or a similar immune system disorder
* Subject does not agree to refrain from any other type of facial skin resurfacing (e.g., microdermabrasion, laser or IPL treatment, chemical peel) or injected filler/other substances (e.g., Restylane, Botox) that might affect the treatment area for the duration of the study
* Underlying silicone or other nonabsorbable fillers in the treatment area or has had filler (e.g., collagen, fat) injections within the past 3 months
* History of keloidal scarring or nodulocystic acne
* Phenol or chemical peel or dermabrasion to the the treatment area within the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Global Acne Scarring Classification | 3 Months post final treatment

SECONDARY OUTCOMES:
Subject Satisfaction | 3 Months post final treatment
  5 point Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Niwat Polnikorn, MD, Principal Investigator — Kasemrad Aesthetic Center, Thailand
Locations (1):
- Kasemrad Aesthetic Center, Kasemrad Prachacheun Hospital, Bangkok, Thailand